CLINICAL TRIAL: NCT06800235
Title: The Effect of Computer-Assisted Simulation Education on Aspiration Skills and General Efficacy Beliefs of Nursing Students
Brief Title: The Effect of Computer-Aided Simulation Training on Aspiration Skills and General Efficacy Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 635
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Aspiration Skill Self-assessment; General Competence Belief
Keywords: aspiration skill self-assessment; general competence belief; computer-based simulation; nursing practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Procedure) (Other): Nursing students in the control group were informed about the standard procedure/traditional method. They were also informed about the aspiration skill form and general competency scale.
  Interventions: Other: Control grup
- Experimental Group (Experimental): Nursing students in the experimental group were informed about computer-based simulation. They were also informed about the aspiration skill form and general competency scale.
  Interventions: Other: Computer-Assisted Simulation

INTERVENTIONS:
Other: Computer-Assisted Simulation — Nursing students in the experimental group were informed about computer-based simulation. They were also informed about the aspiration skill form and general competency scale.
  Arms: Experimental Group
Other: Control grup — Nursing students in the control group were informed about the standard procedure/traditional method. They were also informed about the aspiration skill form and general competency scale.
  Arms: Control Group (Standard Procedure)

SUMMARY:
Purpose This study was conducted to determine the effect of computer-aided simulation education on nursing students' aspiration skills and general competence beliefs.

Research Hypotheses H1-1: Computer-aided simulation education has an effect on aspiration self-efficacy.

H1-2: Computer-aided simulation education has an effect on nursing students' general competence beliefs.

Method

Research Design The research is a randomized controlled experimental study.

Place of the Research The research was conducted with students studying in the second year of the nursing department of the faculty of health sciences of a state university in the fall semester of the 2024-2025 academic year between November 20 and December 20, 2024.

The Universe and Sample of the Study The universe of the study consisted of students studying in the second year of the nursing department of the faculty of health sciences of a state university in the fall semester of the 2024-2025 academic year (N=126). The sample consisted of second year students who met the acceptance criteria of the study. Power analysis was performed to determine the number of people to be included in the study. Power analysis was calculated with the G*Power 3.1 program in the sample calculation. The effect size was taken as 0.80 as high level according to the difference between independent groups determined by Cohen (1988). In order to exceed the 95% value in determining the power of the study; a total of 70 people should be reached, 35 in each group at a significance level of 5% and an effect size of 0.80 (df=68; t=1.668).

The students were randomly assigned to the control and intervention groups. A randomization table was created using the website http://stattrek.com/statistics/random-number-generator.aspx.

DETAILED DESCRIPTION:
Purpose This study was conducted to determine the effect of computer-aided simulation education on nursing students' aspiration skills and general competence beliefs.

Research Hypotheses H1-1: Computer-aided simulation education has an effect on aspiration self-efficacy.

H1-2: Computer-aided simulation education has an effect on nursing students' general competence beliefs.

Method

Research Design The research is a randomized controlled experimental study.

Place of the Research The research was conducted with students studying in the second year of the nursing department of the faculty of health sciences of a state university in the fall semester of the 2024-2025 academic year between November 20 and December 20, 2024.

The Universe and Sample of the Study The universe of the study consisted of students studying in the second year of the nursing department of the faculty of health sciences of a state university in the fall semester of the 2024-2025 academic year (N=126). The sample consisted of second year students who met the acceptance criteria of the study. Power analysis was performed to determine the number of people to be included in the study. Power analysis was calculated with the G*Power 3.1 program in the sample calculation. The effect size was taken as 0.80 as high level according to the difference between independent groups determined by Cohen (1988). In order to exceed the 95% value in determining the power of the study; a total of 70 people should be reached, 35 in each group at a significance level of 5% and an effect size of 0.80 (df=68; t=1.668).

The students were randomly assigned to the control and intervention groups. A randomization table was created using the website http://stattrek.com/statistics/random-number-generator.aspx. Inclusion and Exclusion Criteria: Volunteer second-year nursing students were included in the study. Students who were absent from classes in the relevant period, who joined the department through horizontal and vertical transfer, who were unsuccessful in the Fundamentals of Nursing course, who experienced aspiration skill on a real patient, and students who did not volunteer to participate in the study will not be accepted.

Dependent, independent variables: The dependent variables of the study were determined as aspiration self-efficacy and general competence belief scale score average. Independent variables are other characteristics obtained in the student identification form (age, gender, etc.) Data Collection Tools Student Identification Form It was prepared by the researchers in line with the literature. It consists of 6 questions that include the introductory characteristics of nursing students and some information about their education (age, gender, academic grade point average, type of high school graduated, status of choosing the nursing department, status of fear of performing nursing practices).

Aspiration Skill Self-Assessment Form It was created by the researcher in order to evaluate the students' ability to perform the steps of the procedure related to aspiration application. The first form consisting of 25 items in a 5-point Likert type developed by the researchers for aspiration application skills was presented to a total of 10 experts from the field of nursing. The content validity index (CVI) of the expressions for the created items was calculated. In line with the expert opinions; adjustments were made regarding the items that were stated to be incomprehensible, had similar meanings, contained multiple judgments and would not measure the skill. In addition, the Cronbach Alpha value of the evaluation form for this study was determined as 0.882.

General Competence Belief Scale The scale to be used to measure the general competence belief of nursing students was created by Jerusalem and Schwarzer in 1992. Its adaptation to Turkish was also made by Çelik Kaleli and Çapri (2008) (Çelik Kaleli and Çapri, 2008). The scale has 10 items and a 4-point Likert type. The minimum score that can be obtained from the scale is 10, and the maximum score is 40. An increase in the score obtained by the participant indicates that the level of general competence belief also increases. The Cronbach Alpha value of the scale is 0.92. The Cronbach Alpha value of the scale for this study was obtained as 0.875.

Data Collection The data were collected by the researchers between November-December 2024. The study was started after obtaining permission from the ethics committee and the institution. At the beginning of the study, the purpose and process of the study were explained to the students and the "Informed Voluntary Consent Form" and "Student Identification Form" were filled out. After this consent, other forms were applied to the students as a pre-test. Then, the students were separated into experimental and control groups with a random number table and the education date and information were shared with the students. In the study, the control group was given standard education with a skill model and the experimental group was given education with a computer-aided simulation. The forms were applied again as a post-test after each group.

Ethical Aspect of the Study Before starting the study, approval was obtained from the Istanbul Beykent University Non-Interventional Ethics Committee (Date: 18.11.2024 and Number: 72128186/635) and institutional permission was obtained from the Tekirdağ Namık Kemal University Faculty of Health Sciences. The students were informed about the study and written consent was obtained from the students who volunteered to participate in the study. The study was conducted according to the principles of the Helsinki Declaration.

Data Evaluation The data obtained in the study were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods were used in the evaluation of the data: number, percentage, mean, standard deviation. Differences between the rates of categorical variables in independent groups were analyzed with Chi-Square and Fisher exact tests. Independent groups t-test was used to compare quantitative continuous data between two independent groups. Dependent groups t-test was used to compare within-group measurements. The results were evaluated at a 95% confidence interval and significance was at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Participants;

* Must be enrolled in a nursing program,
* Must be a second year student,
* Must be volunteers for the study.

Exclusion Criteria:

Participants;

* Not registered in the nursing program,
* Not being a second year student,
* Having class absences,
* Joining the department through horizontal or vertical transfer,
* Not passing the Fundamentals of Nursing course,
* Not having experienced aspiration skills on a real patient,
* Not volunteering for the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Aspiration Skill Self-Assessment score average | 1 month
  Nursing students were informed about the Aspiration Skill Self-Assessment Form
General Self-Efficacy Belief Scale score average | 1 month
  Nursing students were informed about the general competency scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, Phd RN, Principal Investigator — Istanbul Beykent University
Locations (1):
- Hamiyet Kızıl, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gülbetekin, E., & Abi, Ö. (2023). Hemşirelik öğrencilerinin mesleki beceri laboratuvarı uygulamaları öncesi ve sonrası stres ve genel yetkinlik inancı düzeyleri: Hemşirelik öğrencilerinin mesleki beceri laboratuvarı uygulamaları. Journal of Infant, Child and Adolescent Health, 3(2), 111-119.